CLINICAL TRIAL: NCT04072393
Title: A Pilot Trial of Cardiac Rehabilitation for Patients Receiving Radiation Therapy for Thoracic Cancers
Brief Title: Cardiac Rehabilitation for Patients Receiving Radiation Therapy for Thoracic Cancers
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Futility
Sponsor: Washington University School of Medicine (Other)
Collaborators: The Foundation for Barnes-Jewish Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 201909133
Record Dates: First submitted 2019-08-26; First posted 2019-08-28 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Lung Cancer; Esophageal Cancer; Thoracic Cancer; Hodgkin Lymphoma; Hodgkin Disease; Non-hodgkin Lymphoma; Sarcoma; Thymoma; Breast Cancer
MeSH Terms: conditions — Lung Neoplasms; Esophageal Neoplasms; Hodgkin Disease; Lymphoma, Non-Hodgkin; Sarcoma; Thymoma; Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Home-based cardiac rehabilitation (Experimental): * The intervention consists of a prescribed course of home-based cardiac rehabilitation: 36 sessions, three times a week, one hour each, over a period of 12 weeks.
  * Each customized exercise session includes three phases:
    * a 5- to 10-minute warm-up which consists of stretching, flexibility movements, and aerobic activity which gradually raises the heart rate to the desired level
    * a conditioning or training phase, which consists of 20 to 45 minutes of continuous or discontinuous aerobic activity
    * a cool down for 5 to 10 minutes consisting of low-intensity exercise that permits a gradual recovery from the conditioning phase
  * The patient will complete a brief questionnaire on the teleHeart application after completing each exercise session on how well they tolerated the exercise. The patient's CR team will receive daily updates from the patient's teleHeart application. Based on feedback from the application, the CR team may modify the patient's exercise program going forward.
  Interventions: Procedure: Home-based cardiac rehabilitation

INTERVENTIONS:
Procedure: Home-based cardiac rehabilitation — -Patients will be evaluated by the clinical team at The Heart Care Institute (HCI). They will receive a heart rate monitor, blood pressure monitor, and weight scale that they will take home with them. They will receive training on how to use the heart rate monitor and blood pressure monitor. They will receive training on how to record their exercises and weights in the teleHeart application by an exercise physiologist from HCI. Within 6 weeks of completion of standard of care radiation therapy or cytotoxic chemotherapy (whichever is last), they will be prescribed a course of home-based CR by a cardiologist at HCI and be instructed on the regimen by an exercise physiologist from HCI.

SUMMARY:
Other than optimizing medical management of cardiac risk factors, and reducing radiotherapy (RT) dose to the heart, there currently exist no interventions to mitigate or reverse the adverse cardiac effects of RT. Aerobic exercise has been demonstrated to improve patient quality of life, cardiac outcomes, and cardiorespiratory fitness in patients with cancer receiving cardiotoxic systemic therapies, but the effects of aerobic exercise on patients at high risk for radiation induced heart disease (RIHD) is unknown. In addition, home-based cardiac rehabilitation has not been tested in patients with thoracic cancers.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed or radiographically diagnosed non-small cell lung cancer, small cell lung cancer, esophageal cancer, Hodgkin lymphoma, non-Hodgkin lymphoma, sarcoma, thymoma, or left-sided breast cancer.
* Planning to receive neo-adjuvant, adjuvant, or definitive radiation therapy to the thorax with curative intent.
* Willing to participate in home-based cardiac rehabilitation program and be monitored remotely via smart phone application
* Possess a smart phone or tablet capable of supporting teleHeart application
* Willing and eligible to co-enroll in the Cardiovascular Toxicity in Cancer and Improvement in Recovery (SURVIVE) Registry Study (HRPO# 201801031).
* At least 18 years of age.
* ECOG performance status ≤ 2
* Ability to understand and willingness to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).

Exclusion Criteria:

* Presence of distant metastatic disease (except patients with lymphoma).
* Life expectancy less than 6 months
* Patient lives in skilled nursing facility, chronic care facility, nursing home, or palliative care or hospice facility
* Unable to walk
* Presence of significant cancer disease burden that would make patient unlikely to tolerate cardiac rehabilitation (CR)
* Diagnosis of primary cervical esophageal cancer.
* Presence of unstable angina.
* Recipient of heart transplant.
* Patient on cardiac transplant list or has a ventricular assist device
* Patient's baseline weight > 300 lbs (due to weight limitations of the scale and bioelectrical impedance device)
* Pregnant and/or breastfeeding. Women of childbearing potential must have a negative pregnancy test within 14 days of study entry.
* Other medical comorbidities that make the patient unable to participate in the CR program or other assessments involved with this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-05-15 (Actual)

PRIMARY OUTCOMES:
Feasibility of completing home-based CR after definitive radiation therapy in patients with thoracic cancer who have started the CR program | Through completion of cardiac rehabilitation for all patients enrolled (estimated to be 36 months)
  Feasibility of completion is defined as 75% of patients who start their first session of cardiac rehabilitation participating in at least 75% of prescribed home-based CR exercise sessions.

SECONDARY OUTCOMES:
Feasibility of home-based cardiac rehabiliation in all enrolled patients after definitive radiation therapy in patients with thoracic cancer. | Through completion of cardiac rehabilitation for all patients enrolled (estimated to be 36 months)
  Feasibility is defined as 75% of all enrolled patients of cardiac rehabilitation participating in at least 75% of prescribed home-based CR sessions.

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Bergom, M.D., Ph.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu